CLINICAL TRIAL: NCT03498508
Title: Poor Theoretical Knowledge and Self-assessed Ability of Cardiopulmonary Resuscitation Among In-hospital Healthcare Professionals: a Cross Sectional Study With Questionnaires.
Status: Completed | Type: Observational
Sponsor: Dalarna County Council, Sweden (Other)
Collaborators: Dalarna University (Other); Center for Clinical Research Dalarna, Sweden (Other); Region Västmanland (Other)
Responsible Party: Principal Investigator, Jennie Silverplats, R.N. PhD candidate, Dalarna County Council, Sweden
Other Study IDs: 2006/201/2 (part 1)
Record Dates: First submitted 2018-03-28; First posted 2018-04-13 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: In-hospital Cardiac Arrest
Keywords: Cardiopulmonary Resuscitation; Knowledge; In-hospital cardiac arrest; Skills

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare professionals in Dalarna County Council: Healthcare professionals working in-hospital at the hospitals in Mora, Avesta and Falun, Sweden, n=1473.
- Healthcare professionals in Region Västmanland: Healthcare professionals working in-hospital at the hospital in Västerås, Region Västmanland, Sweden, n=1571.

SUMMARY:
Theoretical knowledge of cardiopulmonary resuscitation (CPR) is the foundation of being able to perform CPR in a cardiac arrest situation. The knowledge and skills received in training is easily lost and after one year the level is equal to pretraining. International studies regarding knowledge of CPR among healthcare professionals, mostly nurses, show poor results. The knowledge of CPR among Swedish healthcare professionals is poorly studied.

The aim of this study was to describe the theoretical knowledge of CPR and self-assessed abilities of performing CPR among healthcare professionals working in four hospitals in Sweden.

DETAILED DESCRIPTION:
A questionnaire will be handed out containing a knowledge test of nine questions at a basic level. The questionnaire also contains Likert-scales that measures four self-assessed CPR abilities of the respondents (the ability to take leadership, give compressions, to ventilate and to defibrillate).

ELIGIBILITY:
Inclusion Criteria:

* Healtchare professionals of all professions
* Working in-hospital with patient contact
* Present at the time of the survey

Exclusion Criteria:

* Not working with patients
* Abscent at the time of the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare professionals of all professions working in-hospital with patient contact.
Sampling Method: Non-Probability Sample
Enrollment: 3044 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Factors affecting theorethical knowledge | April 30, 2018
  The number of correct answers of the knowledge questions among 3044 respondents will be described and analyzed. An acceptable amount of correct answers will be seven out of nine, or more, >80%. The dependent variable number of correct answers will be analyzed with the independent variables profession, years in profession, workplace and time since last CPR-training.
Factors affecting self-assessed abilities. | April 30, 2018
  Four self-assessed CPR-skills among 3044 respondents measured on a Likert scale of 1-7 will be measured and described. The skills are the ability to take leadership, give chest compressions, to ventilate and to defibrillate. The dependent variable consisting of a factor score of self-assessed abilities will be analyzed with independent variables such as profession, years in profession, workplace and time since last CPR-training.

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Strömsöe, Study Director — Dalarna County Council
Locations (4):
- Sweden (4):
  - Avesta Lasarett, Avesta, Dalarna County
  - Falu Lasarett, Falun, Dalarna County
  - Mora Lasarett, Mora, Dalarna County
  - Västmanlands sjukhus, Västerås, Västmanland County